CLINICAL TRIAL: NCT04773964
Title: Phase 2a Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MET642 in Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Study to Evaluate MET642 in Patients With NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metacrine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MET642-201
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2021-09

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: NASH; Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MET642 high dose (Experimental)
  Interventions: Drug: MET642
- MET642 low dose (Experimental)
  Interventions: Drug: MET642
- MET642 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MET642 — MET642 active treatment
  Arms: MET642 high dose; MET642 low dose
Drug: Placebo — Placebo comparator
  Arms: MET642 Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled study to evaluate MET642 in NASH patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NASH via biopsy, magnetic resonance elastography (MRE), or transient elastography (TE, FibroScan)
* Liver fat content ≥ 10% as measured by magnetic resonance imaging-proton density fat fraction (MRI-PDFF).

Exclusion Criteria:

* History of significant liver disease (eg, alcoholic liver disease, viral hepatitis, etc.) or liver transplant.
* Presence of cirrhosis on any prior liver biopsy (stage 4 fibrosis).
* Excessive consumption of alcohol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 28 days after last dose
  Incidences of treatment-emergent adverse events
Vital Signs | Up to 28 days after last dose
  Incidences of clinically significant changes in vital signs
Laboratory tests | Up to 28 days after last dose
  Incidences of clinically significant changes in laboratory tests
ECG | Up to 28 days after last dose
  Incidences of clinically significant changes in ECGs

SECONDARY OUTCOMES:
Pharmacokinetic Profile of MET642 | 16 weeks
  Cmax
Pharmacodynamic Profile of MET642 | 16 weeks
  C4 concentrations
Pharmacological Activity of MET642 | 20 weeks
  Measure of changes in liver fat using MRI-PDFF
Pharmacokinetic Profile of MET642 | 16 weeks
  Tmax
Pharmacokinetic Profile of MET642 | 16 weeks
  T1/2
Pharmacokinetic Profile of MET642 | 16 weeks
  AUC0-inf
Pharmacodynamic Profile of MET642 | 16 weeks
  FGF19 concentrations
Pharmacodynamic Profile of MET642 | 16 weeks
  Bile Acids concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Pinnacle Research, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Metacrine website — http://www.metacrine.com
- See also: Study website — http://www.nashfxr.com